CLINICAL TRIAL: NCT02806934
Title: Tumor Necrosis Factor-308 Polymorphism a Embryo Implantation Rate in Women Undergoing in Vitro Fertilization
Brief Title: TNF Polymorphism and Implantation Rate
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 08-API-01
Record Dates: First submitted 2016-05-27; First posted 2016-06-21 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Biological Products; High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: biological and ultrasound test — biological and ultrasound test 20 days after implantation in order to see the implantation rate

SUMMARY:
Do TNF-308 and -238 polymorphisms impact the embryo implantation rate after in vitro fertilization (IVF) in women without female infertility factor ?

DETAILED DESCRIPTION:
This study was performed in order to verify whether TNF-308 allele was associated with a higher implantation rate and multiple pregnancy rates in women without known infertility factors after ovarian hyperstimulation with exogenous FSH for IVF

ELIGIBILITY:
Inclusion Criteria:

* Women
* normal karyotype,
* age under 38 years
* serum follicle-stimulating hormone (Day-3 FSH) levels below 10 UI/l

Exclusion Criteria:

* age under 18 years

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women undergoing intracytoplasmic sperm injection (ICSI) due to male infertility factors
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2009-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Implantation rate by biological test | 20 days after implantation
Implantation rate by ultrasound test | 20 days after implantation

CONTACTS AND LOCATIONS:
Overall Officials: Patrick FENICHEL, PU-PH, Principal Investigator — service d'Endocrinologie
Locations (1):
- Nice University Hospital, Nice, France